CLINICAL TRIAL: NCT04037033
Title: Forming New Habits: A Feasibility Study on an Intervention to Decrease Sedentary Behaviors in Medically Stable Older Adults
Brief Title: Habit Formation in Older Adults: Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Young Joo Kim, Assistant Professor, East Carolina University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCIRB 19-001365
Record Dates: First submitted 2019-07-24; First posted 2019-07-30 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Older Adults
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: Single group, pre-post design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Everyday Meaningful Activities (EMA) intervention — The EMA intervention will include 6 intervention sessions. At session 1, the interventionist and participant will identify 2 meaningful active lifestyle behavior goals using COPM. Last, an action plan will be created for behavior 1. Participants will be asked to implement the action plan everyday.
  At session 2, the interventionist and participants will review the daily activity log and the action plan.
  At session 3, the interventionist and the participants will review the daily activity log and the action plan.
  At session 4, an action plan will be created for behavior 2. Participants will be asked to implement the action plan for behavior 2 everyday.
  At session 5, the participants and interventionists will discuss the participant's daily activity log and action plan.
  At session 6, the participants and interventionists will discuss the participant's daily activity log and action plan.

SUMMARY:
Sedentary behavior, which is characterized by too much sitting, is an epidemic in the United States. It is estimated that 4 out of every 10 Americans never engage in physical activity, and approximately 60% of an adult's non-sleeping hours are spent in sedentary behaviors. This equates to approximately 9-10 hours per day. As sedentary behavior increases, so do diagnoses of chronic illnesses such as diabetes, hypertension, cardiovascular disease, and kidney disease. Older adults are particularly at risk for sedentary behavior and the related chronic illnesses.

The primary aim of this study is to investigate the feasibility of implementing the EMA intervention with medically stable older adults who are living in the community.

The secondary aims of this study are to investigate the effectiveness of the Everyday Meaningful Activities (EMA) Intervention in forming active lifestyle behavior habits and in decreasing an individual's perceived sedentary time.

This prospective study will examine the ability of medically stable older adults to decrease sedentary behavior by creating new, active lifestyle behavior habits using the Everyday Meaningful Activities intervention. The EMA Intervention is based in Habit Formation Theory. It is an individualized, client-centered intervention that aims to increase adherence to active lifestyle behaviors in older adults' lives. Participants will engage in the EMA Intervention that is designed to create new active lifestyle behavior habits by attaching these new active lifestyle behaviors to currently existing daily routines.

During six intervention sessions over six weeks, participants will select two new active lifestyle behaviors to make habitual and will create action plans to create the habits. The first behavior will be implemented at the first intervention session, and the second behavior will be implemented at the fourth session. The participants will be assessed three times over their 8 to 10-week study participation. Participants should (1) be 65 years of age and older, (2) have intact cognition, (3) have no self-reported physical activity limitations, (4) have a sedentary lifestyle, and (5) have no acute illnesses or unstable medical conditions.

The results of this study may provide evidence for the occupational therapy intervention to decrease sedentary behavior in older adults in the community. The results may also broaden the scope of occupational therapy practice through demonstrating the potential for occupational therapy services in preventive health care.

ELIGIBILITY:
Inclusion Criteria:

* age 65 or older,
* intact cognition as confirmed by the Montreal Cognitive Assessment blind version
* no physical activity restrictions that can be self-reported
* sedentary lifestyle as confirmed by the Rapid Assessment Disuse Index
* live within 20 miles of the College of Allied Health Sciences at ECU
* have access to the internet and/or a telephone for remote intervention sessions

Exclusion Criteria:

* acute or terminal illness
* myocardial infarction in the previous 6 months
* unstable cardiovascular disease
* unstable metabolic disease
* neuromusculoskeletal disorders that severely impact voluntary movement
* limb amputation
* upper or lower extremity fracture in the previous 3 months
* current symptomatic hernia
* current symptomatic hemorrhoids
* cognitive impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Through study completion, an average of 1 year
  The recruitment rate for medically stable older adults in the community for this study
Appropriateness of the Rapid Assessment Disuse Index (RADI) | During screening
  The appropriateness of the Rapid Assessment Disuse Index (RADI) for screening sedentary behavior in older adults over the phone
Appropriateness of the Short Blessed Test | During screening
  the appropriateness of the Short Blessed Test for screening sufficient cognitive ability in older adults over the phone
Appropriateness of video conferencing through WebEx on an iPad | For 6 weeks
  The appropriateness of video conferencing through WebEx on an iPad as an acceptable delivery method of selected intervention sessions
Reliability of participants' subjective reports | For 6 weeks
  The reliability of participants' subjective reports of exact times for performing active lifestyle behaviors

SECONDARY OUTCOMES:
Changes in the Self-Report Habit Index | 1) intervention session 1 at Week 1; 2) intervention session 4 at Week 4, and 3) posttest at Week 7
  The Self-Report Habit Index (SRHI) measures features of habits including repetition, automaticity, and expressing identity. This 12-item assessment assesses the strength of habits by differentiating habit strength from behavior frequency. The participants will choose two active lifestyle behaviors to incorporate into their daily lives. The SRHI will generate pretest and posttest data for each behavior. The items in the SRHI began with the stem "Behavior X is something…" and is then followed by 12 statements rated on a scale from 1 (very strongly agree) to 7 (very strongly disagree). A total score ranges from 1 to 84 with lower scores indicating stronger habits.
Changes in Sedentary Behavior Questionnaire | 1) intervention session 1 at Week 1, and 2) posttest at Week 7
  The Sedentary Behavior Questionnaire (SBQ) is a self-report questionnaire about time spent in sedentary behaviors both on weekdays and weekends. There are 9 identical items on the weekday form and the weekend form. Participants will complete both forms at both time points. The SBQ is used to assess the participants' perceived sedentary time. A total score ranges from 0 to 54 for each (weekday and weekend), with higher scores indicating more sedentary behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Young Joo Kim, PhD, Principal Investigator — East Carolina University
Locations (1):
- East Carolina University, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No